CLINICAL TRIAL: NCT03743558
Title: Screening of Obstructive Sleep Apnea by Smartphone Homemade Video in Childood Snoring Population
Acronym: SMARTSAS
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: difficulty of recrutement
Sponsor: University Hospital, Clermont-Ferrand (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: CHU-414; 2018-A00435-50 (Other: 2018-A00435-50)
Record Dates: First submitted 2018-11-05; First posted 2018-11-16 (Actual); Last update posted 2024-03-07 (Actual); Status verified 2024-03

CONDITIONS: Obstructive Sleep Apnea Syndrome; Adeno-amygdala Hypertrophy; Snoring
Keywords: Obstructive sleep apnea syndrome; Adeno-amygdala hypertrophy; Tonsillectomy; Video; Smartphone; Ventilatory polygraphy
MeSH Terms: conditions — Sleep Apnea, Obstructive; Snoring

STUDY DESIGN:
Intervention Model Description: First consultation: SHS questionnaire submission and clinical examination
  * Realization of PV and analysis according to the standard criteria of the American Academy of Sleep Medicine
  * Production of a video at home by the parents according to the following conditions, within 4 days around the PV/PSG :
  * Second consultation
  * Collection of the video and the result of the PV
  * Study exit.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- children with adenoamygdala hypertrophy (Experimental)
  Interventions: Behavioral: smartphone homemade video

INTERVENTIONS:
Behavioral: smartphone homemade video — value of a video recording of the child sleep on smartphone made by the parents

SUMMARY:
The aim of the study is to evaluate the value of a video recording of the child sleep on smartphone made by the parents and comparing it to ventilatory polygraphy (PV) on the one hand and to the clinical evaluation method (clinical examination + Spruyt and Gozal score) on the other hand.

DETAILED DESCRIPTION:
Obstructive sleep apnoea syndrome (OSAS) is a common disorder in school-aged children with an estimated prevalence of 1-4%. The main etiology is adeno-amygdala hypertrophy. Adenoamygdalectomy, which involves the removal of tonsils and adenoids, is a common procedure. In the majority of cases, it allows the healing of OSAS. The surgical indication is currently based on clinical arguments sensitized by the calculation of a severity score (Spruyt and Gozal score). However, this procedure is not without complications: pneumopathy (for 1.5% of procedures), blood transfusion for haemorrhage (1/400 to 1/2 500), death due to haemorrhage (1/35 000 to 1/50 000).

Currently there is no indication to perform a preoperative sleep recording for this surgery. This recording will only be made in case of associated comorbidities (obesity, craniofacial malformations, neurological disorders...).

The current growth and diffusion of smartphones in the population provides a simple technical means of video recording the child's sleep. More and more parents come to an ENT consultation with a video recording of their child's sleep on a smartphone. The current recommendations say to take these data into account without any study having evaluated the value of such records. The video recording of a snoring child's sleep has already been evaluated by Sivan et al in 1996. This study finds a good correlation between polysomnographic recording and a method of rating video recordings of sleep in children with adeno-amygdala hypertrophy without associated comorbidities.

The aim of this study is therefore to evaluate the value of this video recording on smartphone made by the parents by comparing it to ventilatory polygraphy (PV) on the one hand and to the clinical evaluation method (clinical examination + SHS score) on the other hand. If our hypothesis is correct, smartphone video recording could be an additional tool to the clinical diagnosis of OSA in children with adeno-amygdala hypertrophy.

ELIGIBILITY:
Inclusion Criteria:

* Children between 3 and 10 years old consulting an ENT for snoring noted by the entourage (parents).
* Tonsil hypertrophy ≥ 2 (Brodsky classification).
* Entourage in possession of a smartphone allowing a video recording (under Android format).

Exclusion Criteria:

* Chronic cardiovascular, neurological, metabolic (overweight, obesity) or associated pulmonary pathology.
* Syndromic craniofacial malformations.

Ages: 3 Years to 10 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 56 (Actual)
Dates: Start 2019-02-13 (Actual); Primary Completion 2022-05-11 (Actual); Study Completion 2022-05-11 (Actual)

PRIMARY OUTCOMES:
Video analysis score | at day 1
  The primary judging criterion will be the 10-minute video analysis score (independent variable). The dependent variable will be the status obtained with PV (pathological or normal), defined according to the standard criteria of the American Academy of Sleep Medicine 2012
status obtained with PV | at day 1
  The primary judging criterion will be the 10-minute video analysis score (independent variable). The dependent variable will be the status obtained with PV (pathological or normal), defined according to the standard criteria of the American Academy of Sleep Medicine 2012

SECONDARY OUTCOMES:
Video analysis score | at day 1
  The secondary judging criterion will be the 10-minute video analysis score (independent variable). The dependent variable will be the status obtained with the score from the Spruyt and Gozal questionnaire (hierarchical SHS severity score) in its validated version in French.
score from the Spruyt and Gozal questionnaire | at day 1
  The secondary judging criterion will be the 10-minute video analysis score (independent variable). The dependent variable will be the status obtained with the score from the Spruyt and Gozal questionnaire (hierarchical SHS severity score) in its validated version in French.

CONTACTS AND LOCATIONS:
Overall Officials: Nicolas SAROUL, Principal Investigator — University Hospital, Clermont-Ferrand
Locations (1):
- Chu Clermont-Ferrand, Clermont-Ferrand, France

REFERENCES:
- [Background] Pateron B, Marianowski R, Monteyrol PJ, Couloigner V, Akkari M, Chalumeau F, Fayoux P, Leboulanger N, Franco P, Mondain M. French Society of ENT (SFORL) guidelines (short version) on the roles of the various treatment options in childhood obstructive sleep apnea-hypopnea syndrome. Eur Ann Otorhinolaryngol Head Neck Dis. 2018 Aug;135(4):265-268. doi: 10.1016/j.anorl.2018.04.005. Epub 2018 May 3. PMID 29731297
- [Background] Spruyt K, Gozal D. Screening of pediatric sleep-disordered breathing: a proposed unbiased discriminative set of questions using clinical severity scales. Chest. 2012 Dec;142(6):1508-1515. doi: 10.1378/chest.11-3164. PMID 22677350
- [Background] Nguyen XL, Levy P, Beydon N, Gozal D, Fleury B. Performance characteristics of the French version of the severity hierarchy score for paediatric sleep apnoea screening in clinical settings. Sleep Med. 2017 Feb;30:24-28. doi: 10.1016/j.sleep.2016.01.021. Epub 2016 Mar 14. PMID 28215255
- [Background] Sivan Y, Kornecki A, Schonfeld T. Screening obstructive sleep apnoea syndrome by home videotape recording in children. Eur Respir J. 1996 Oct;9(10):2127-31. doi: 10.1183/09031936.96.09102127. PMID 8902478
- [Background] Berry RB, Budhiraja R, Gottlieb DJ, Gozal D, Iber C, Kapur VK, Marcus CL, Mehra R, Parthasarathy S, Quan SF, Redline S, Strohl KP, Davidson Ward SL, Tangredi MM; American Academy of Sleep Medicine. Rules for scoring respiratory events in sleep: update of the 2007 AASM Manual for the Scoring of Sleep and Associated Events. Deliberations of the Sleep Apnea Definitions Task Force of the American Academy of Sleep Medicine. J Clin Sleep Med. 2012 Oct 15;8(5):597-619. doi: 10.5664/jcsm.2172. PMID 23066376